CLINICAL TRIAL: NCT02605148
Title: TEFA TEDDY Family Prevention - Gluten Free Diet to Preserve Beta-cell Function in Subjects With Islet Autoimmunity.
Brief Title: TEFA Family Prevention: Glutenfree Diet to Preserve Beta-cell Function
Acronym: TEFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lund University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Maria Månsson Martinez, Study coordinator, Lund University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TEFA/2015
Record Dates: First submitted 2015-11-11; First posted 2015-11-16 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Prediabetes; Type 1 Diabetes
Keywords: Islet autoimmunity; gluten free diet; prediabetes; prevention; type 1 diabetes; glucose tolerance test
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 1 | interventions — Diet, Gluten-Free; Fatty Acids, Omega-3; Vitamin D; Probiotics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gluten free diet (Experimental): Gluten free diet during 18 months. The subjects will be referred to a nutritionist every 6 months. Vitamin D 800 U Daily, Omega 3 fatty acids and probiotics as nutritional supplements.
  Interventions: Dietary Supplement: Gluten free diet; Dietary Supplement: Omega 3 fatty acid; Dietary Supplement: Vitamin D; Dietary Supplement: Probiotics
- Normal diet (Active Comparator): Normal diet. Vitamin D 800 U Daily, Omega 3 fatty acids and probiotics as nutritional supplements.
  Interventions: Dietary Supplement: Omega 3 fatty acid; Dietary Supplement: Vitamin D; Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Gluten free diet — Gluten free diet during 18 months.
  Arms: Gluten free diet
Dietary Supplement: Omega 3 fatty acid — Omega 3 fatty acid
Dietary Supplement: Vitamin D — Vitamin D 800 U/day
Dietary Supplement: Probiotics — Probiotics

SUMMARY:
To evaluate the effect of Gluten Free Diet (GFD) on beta-cell function and glucose metabolism in subjects with one or several islet autoantibodies without and with dysglycemia at baseline. Additionally, all subjects will be given treatment with Vitamin D, omega fatty acids and probiotics.

Subjects will be randomized to GFD or normal diet during 18 months. Beta cell function will be evaluated at baseline, and during follow-up by glucose tolerance tests.

DETAILED DESCRIPTION:
The design is a randomized controlled study to determine the safety and the effect of gluten free diet during 18 months on beta-cell function and glucose metabolism. Lead-in and nonstop supplement cocktail including vitamin D, omega fatty acids and probiotics will be used to equalize differences to reduce known confounders. All study subjects will meet with a dietician to obtain a 3-day diet record and to receive instructions on a healthy normal diet or GFD.

Subjects (n=60) at 2-49.99 years of age positive for one or several islet autoantibodies will be recruited. Subjects with one islet autoantibody have done one or several oral glucose tolerance test (OGTT) prior to the baseline visit. One islet autoantibody positive subjects are only eligible if they have dysglycemia. All subjects will be randomized based on baseline intravenous glucose tolerance test (IvGTT) and OGTT into subjects without and with dysglycemia at baseline.

Beta-cell function and glucose metabolism (alternating IvGTT and OGTT) will be assessed at baseline and after 6, 12, 18 months of treatment and after 6 months of wash out on a normal healthy diet.

Adverse events and safety Adverse event will be obtained at visits and during the study, which will be monitored.

It is expected that subjects with one or several islet autoantibodies will show a loss compared to baseline of beta-cell function and glucose control. GFD is expected to reduce the loss in subjects on a healthy diet.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects from two (2) to 49,99 years of age.
2. At least one type 1 diabetes-associated autoantibody (to glutamic acid (GADA), insulin (IAA), insulinoma-associated protein 2 (IA-2A) or zinktransporter 8 (ZnT8R/W/QA) in subjects with impaired glucose metabolism OR at least two type 1 diabetes-associated autoantibodies, regardless of normal or impaired glucose metabolism.
3. Written informed consent from research subject. If a child, also from the child's parents or legal acceptable representative(s) according to local regulations.

Exclusion Criteria:

1. Ongoing treatment with immunosuppressant therapy (topical or inhaled steroids are accepted).
2. Diabetes.
3. Treatment with any oral or injected anti-diabetic medications.
4. Significantly abnormal hematology results at screening.
5. Participation in other clinical trials with a new chemical entity within the previous 3 months.
6. History of hypercalcemia.
7. Presence of associated serious disease or condition.
8. Diabetes-protective HLA-DQ6-allele.

   -

Ages: 2 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-12; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in first phase insulin response (FPIR) from IvGTT | 24 months
  Change in First phase insulin response from IvGTT during follow-up
Change in area under the curve (AUC) C-peptide | 24 months
  Change in AUC C-peptide from OGTT during follow-up
Change in glucose metabolism | 24 months
  Change from normal to impaired glucose metabolism during follow-up

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 24 months
  To evaluate safety of GFD compared to recommended normal diet in the placebo group in subjects supplemented with lead in and nonstop treatment with a cocktail including vitamin D, omega fatty acids and probiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Månsson Martinez, Nutricionist, Principal Investigator — Lund University
Locations (1):
- Lund University, Department of Clinical Sciences Malmö, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez MM, Spiliopoulos L, Salami F, Agardh D, Toppari J, Lernmark A, Kero J, Veijola R, Tossavainen P, Palmu S, Lundgren M, Borg H, Katsarou A, Larsson HE, Knip M, Maziarz M, Torn C; and the TEDDY-Family (TEFA) Study Group. Heterogeneity of beta-cell function in subjects with multiple islet autoantibodies in the TEDDY family prevention study - TEFA. Clin Diabetes Endocrinol. 2022 Jan 5;7(1):23. doi: 10.1186/s40842-021-00135-6. PMID 34983671
- [Derived] Martinez MM, Salami F, Larsson HE, Toppari J, Lernmark A, Kero J, Veijola R, Koskenniemi JJ, Tossavainen P, Lundgren M, Borg H, Katsarou A, Maziarz M, Torn C; TEDDY Family (TEFA) Study Group. Beta cell function in participants with single or multiple islet autoantibodies at baseline in the TEDDY Family Prevention Study: TEFA. Endocrinol Diabetes Metab. 2020 Nov 5;4(2):e00198. doi: 10.1002/edm2.198. eCollection 2021 Apr. PMID 33855205